CLINICAL TRIAL: NCT01962415
Title: A Phase II Study of Reduced Intensity Conditioning in Pediatric Patients and Young Adults ≤55 Years of Age With Non-Malignant Disorders Undergoing Umbilical Cord Blood, Bone Marrow, or Peripheral Blood Stem Cell Transplantation
Brief Title: Reduced Intensity Conditioning for Non-Malignant Disorders Undergoing UCBT, BMT or PBSCT
Acronym: HSCT+RIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, BMT-CT at CHP of UPMC and Professor of Pediatrics and Immunology, University of Pittsburgh, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19060337
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Primary Immunodeficiency (PID); Congenital Bone Marrow Failure Syndromes; Inherited Metabolic Disorders (IMD); Hereditary Anemias; Inflammatory Conditions; Systemic Juvenile Idiopathic Arthritis (sJIA); Juvenile Rheumatoid Arthritis (JRA)
Keywords: Severe Combined Immune Deficiency (SCID); Omenn Syndrome; Bare Lymphocyte Syndrome (BLS); Combined Immune Deficiency (CID) syndromes; Combined Variable Immune Deficiency (CVID) syndrome; Wiskott-Aldrich Syndrome; Leukocyte adhesion deficiency; Chronic granulomatous disease (CGD); X-linked Hyper IgM (XHIM) syndrome; IPEX syndrome; Chediak - Higashi Syndrome; Autoimmune Lymphoproliferative Syndrome (ALPS); Hemophagocytic Lymphohistiocytosis (HLH) syndromes; Lymphocyte Signaling defects; Dyskeratosis Congenita (DC); Congenital Amegakaryocytic Thrombocytopenia (CAMT); Osteopetrosis; Mucopolysaccharidoses; Hurler syndrome (MPS I); Hunter syndrome (MPS II); Leukodystrophies; Krabbe Disease; Metachromatic leukodystrophy (MLD); X-linked adrenoleukodystrophy (ALD); Alpha mannosidosis; Gaucher Disease; Thalassemia major; Sickle cell disease (SCD); Diamond Blackfan Anemia (DBA); Crohn's Disease; Inflammatory Bowel Disease; Hematopoietic Stem Cell Transplant (HSCT); Congenital transfusion dependent anemias; Globoid cell leukodystrophy; Hereditary diffuse leukoencephalopathy with spheroids (HDLS); Systemic Juvenile Idiopathic Arthritis (sJIA); Juvenile Rheumatoid Arthritis (JRA)
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Congenital Bone Marrow Failure Syndromes; Arthritis, Juvenile; Severe Combined Immunodeficiency; Syndrome; Wiskott-Aldrich Syndrome; Leukocyte adhesion deficiency type 1; Granulomatous Disease, Chronic; Immune Dysregulation, Polyendocrinopathy, Enteropathy, X-Linked Syndrome; Chediak-Higashi Syndrome; Autoimmune Lymphoproliferative Syndrome; Lymphohistiocytosis, Hemophagocytic; Dyskeratosis Congenita; Congenital amegakaryocytic thrombocytopenia; Osteopetrosis; Mucopolysaccharidoses; Mucopolysaccharidosis I; Mucopolysaccharidosis II; Sudden Infant Death; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Adrenoleukodystrophy; alpha-Mannosidosis; Gaucher Disease; beta-Thalassemia; Anemia, Sickle Cell; Anemia, Diamond-Blackfan; Crohn Disease; Inflammatory Bowel Diseases; Hereditary Diffuse Leukoencephalopathy with Spheroids | interventions — Hydroxyurea; Alemtuzumab; fludarabine; fludarabine phosphate; Melphalan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- UCBT:transfusion dependent anemias or increased rejection risk (Experimental): Alemtuzumab, Hydroxyurea, Fludarabine, Melphalan, and Thiotepa conditioning regimen prior to allogenic HSCT.
  Interventions: Drug: Hydroxyurea; Drug: Alemtuzumab; Drug: Fludarabine; Drug: Melphalan; Drug: Thiotepa
- BMT, PBSCT and not transfusion dependent UCBT (Experimental): Alemtuzumab, Hydroxyurea, Fludarabine, Melphalan, and Thiotepa conditioning regimen prior to allogenic HSCT.
  Interventions: Drug: Hydroxyurea; Drug: Alemtuzumab; Drug: Fludarabine; Drug: Melphalan; Drug: Thiotepa

INTERVENTIONS:
Drug: Hydroxyurea — Oral administration
  Other Names: hydroxycarbamide; Hydrea; Droxia
Drug: Alemtuzumab — Intravenous (IV) administration.
  Other Names: Campath
Drug: Fludarabine — IV administration
  Other Names: Fludara
Drug: Melphalan — IV administration
  Other Names: Melphalan hydrochloride; Alkeran
Drug: Thiotepa — IV administration

SUMMARY:
The objective of this study is to evaluate the efficacy of using a reduced-intensity condition (RIC) regimen with umbilical cord blood transplant (UCBT), double cord UCBT, matched unrelated donor (MUD) bone marrow transplant (BMT) or peripheral blood stem cell transplant (PBSCT) in patients with non-malignant disorders that are amenable to treatment with hematopoietic stem cell transplant (HSCT). After transplant, subjects will be followed for late effects and for ongoing graft success.

DETAILED DESCRIPTION:
For some non-malignant diseases (NMD; i.e., thalassemia, sickle cell disease, most immune deficiencies) a hematopoietic stem cell transplant may be curative by healthy donor stem cell engraftment alone. HSCT in patients with NMD differs from that in malignant disorders for two important reasons: 1) these patients are typically naïve to chemotherapy and immunosuppression. This may potentially lead to difficulties with engraftment. And 2) RIC with subsequent bone marrow chimerism may be beneficial even in mixed chimerism and result in decreased transplant-related mortality (TRM). Nevertheless, any previous organ damage, as a result of the underlying disease, may remain present after the HSCT.

For other diseases (metabolic disorders, some immunodeficiencies, etc.), a transplant is not curative. For these diseases, the main intent of the transplant is to slow down, or stop, the progress of the disease. In select few cases/diseases, the presence of healthy bone marrow derived cells may even prevent progression and prevent neurological decline.

Research funds are not available to assist with enrollment on this trial.

In this research study, instead of using the standard myeloablative conditioning, the study doctor is using RIC, in which significantly lower doses of chemotherapy will be used. The lower doses may not eradicate every stem cell in the patient's bone marrow, however, in the presented combination, the intention is to eliminate already formed immune cells and provide maximum growth advantage to healthy donor stem cells. This paves the way to successful engraftment of donor stem cells. Engrafting donor stem cells can outcompete, and donor lymphocytes could suppress, the patients' surviving stem cells. With RIC, the side effects on the brain, heart, lung, liver, and other organ functions are less severe and late toxic effects should also be reduced.

The purpose of this study is to collect data from the patients undergoing reduced-intensity conditioning before HSCT, and compare it to the standard myeloablative conditioning. It is expected there will be therapeutic benefits, paired with better survival rate, less organ toxicity and improved quality of life, following the RIC compared to the myeloablative regimen.

ELIGIBILITY:
Inclusion:

1. A 4/6, 5/6 or 6/6 HLA matched related or unrelated UCB unit available that will deliver a pre-cryopreservation total nucleated cell dose of ≥ 3 x 10e7 cells/kg, or double unit grafts, each cord blood unit delivering at least 2 x 10e7 cells/kg OR an 8 of 8 or 7 of 8 HLA allele level matched unrelated donor bone marrow or peripheral blood progenitor graft.
2. Adequate organ function as measured by:

   1. Creatinine ≤ 2.0 mg/dL and creatinine clearance ≥ 50 mL/min/1.73 m2.
   2. Hepatic transaminases (ALT/AST) ≤ 4 x upper limit of normal (ULN).
   3. Adequate cardiac function by echocardiogram or radionuclide scan (shortening fraction > 26% or ejection fraction > 40% or > 80% of normal value for age).
   4. Pulmonary evaluation testing demonstrating CVC or FEV1/FVC of ≥ 50% of predicted for age and/or resting pulse oximeter ≥ 92% on room air or clearance by the pediatric or adult pulmonologist. For adult patients DLCO (corrected for hemoglobin) should be ≥ 50% of predicted if the DLCO can be obtained.
3. Written informed consent and/or assent according to FDA guidelines.
4. Negative pregnancy test if pubertal and/or menstruating.
5. HIV negative.
6. A non-malignant disorder amenable to treatment by stem cell transplantation, including but not limited to:

   1. Primary Immunodeficiency syndromes including but not limited to:

      * Severe Combined Immune Deficiency (SCID) with NK cell activity
      * Omenn Syndrome
      * Bare Lymphocyte Syndrome (BLS)
      * Combined Immune Deficiency (CID) syndromes
      * Combined Variable Immune Deficiency (CVID) syndrome
      * Wiskott-Aldrich Syndrome
      * Leukocyte adhesion deficiency
      * Chronic granulomatous disease (CGD)
      * X-linked Hyper IgM (XHIM) syndrome
      * IPEX syndrome
      * Chediak - Higashi Syndrome
      * Autoimmune Lymphoproliferative Syndrome (ALPS)
      * Hemophagocytic Lymphohistiocytosis (HLH) syndromes
      * Lymphocyte Signaling defects
      * Other primary immune defects where hematopoietic stem cell transplantation may be beneficial
   2. Congenital bone marrow failure syndromes including but not limited to:

      * Dyskeratosis Congenita (DC)
      * Congenital Amegakaryocytic Thrombocytopenia (CAMT)
      * Osteopetrosis
   3. Inherited Metabolic Disorders (IMD) including but not limited to:

      * Mucopolysaccharidoses

        * Hurler syndrome (MPS I)
        * Hunter syndrome (MPS II)
      * Leukodystrophies

        * Krabbe Disease, also known as globoid cell leukodystrophy
        * Metachromatic leukodystrophy (MLD)
        * X-linked adrenoleukodystrophy (ALD)
        * Hereditary diffuse leukoencephalopathy with spheroids (HDLS)
      * Other inherited metabolic disorders

        * alpha mannosidosis
        * Gaucher Disease
      * Other inheritable metabolic diseases where hematopoietic stem cell transplantation may be beneficial.
   4. Hereditary anemias

      * Thalassemia major
      * Sickle cell disease (SCD) - patients with sickle disease must have one or more of the following:

        * Overt or silent stroke
        * Pain crises ≥ 2 episodes per year for past year
        * One or more episodes of acute chest syndrome
        * Osteonecrosis involving ≥ 1 joints
        * Priapism
      * Diamond Blackfan Anemia (DBA)
      * Other congenital transfusion dependent anemias
   5. Inflammatory Conditions

      * Crohn's Disease/Inflammatory Bowel Disease

Exclusion:

1. Allogeneic hematopoietic stem cell transplant within the previous 6 months.
2. Any active malignancy or MDS.
3. Severe acquired aplastic anemia.
4. Uncontrolled bacterial, viral or fungal infection (currently taking medication and with progression of clinical symptoms).
5. Pregnancy or nursing mother.
6. Poorly controlled pulmonary hypertension.
7. Any condition that precludes serial follow-up.

Ages: 2 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-02-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Post-transplant treatment-related mortality (TRM) | 1 year post-transplant
  The number of deaths related to the research intervention at day 100, 6 months, and 1 year post-transplant.
Neurodevelopmental milestones | 1 year post-transplant
  Evaluation of the pace of attaining neurodevelopmental milestones after reduced-intensity conditioning as compared to myeloablative conditioning historical controls from the target population(s).
Immune Reconstitution | 1 year post-transplant
  Evaluation of the pace of immune reconstitution.
Severe opportunistic infections | 1 year post-transplant
  Evaluation of the incidence of severe opportunistic infections.
GVHD occurrence | 1 year post-transplant
  Description of the incidence of acute graft versus host disease (GVHD) (II-IV) and chronic extensive GVHD.

SECONDARY OUTCOMES:
Donor cell engraftment | 6 months post-transplant
  Determination of the feasibility of attaining robust donor cell engraftment (>50% donor chimerism at 6 months) following reduced-intensity conditioning (RIC) regimens prior to HSCT in the target population(s).
Normal enzyme level | 1 year post-transplant
  Determination of the feasibility of attaining and sustaining normal enzyme levels in the target population(s).
Neutrophil recovery | 1 year post-transplant
  Determination of the pace of neutrophil recovery.
Platelet recovery | 1 year post-transplant
  Determination of the pace of platelet recovery.
Grade 3-4 organ toxicity | 1 year post-transplant
  The number of grade 3-4 organ adverse events.
Late graft failure | 1 year post-transplant
  Evaluation of the incidence of late graft failure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vander Lugt MT, Chen X, Escolar ML, et al. Reduced-intensity single-unit unrelated cord blood transplant with optional immune boost for nonmalignant disorders. Blood Adv. 2020;4(13):3041-3052. Blood Adv. 2020 Aug 11;4(15):3508. doi: 10.1182/bloodadvances.2020002967. No abstract available. PMID 32750127
- [Derived] Vander Lugt MT, Chen X, Escolar ML, Carella BA, Barnum JL, Windreich RM, Hill MJ, Poe M, Marsh RA, Stanczak H, Stenger EO, Szabolcs P. Reduced-intensity single-unit unrelated cord blood transplant with optional immune boost for nonmalignant disorders. Blood Adv. 2020 Jul 14;4(13):3041-3052. doi: 10.1182/bloodadvances.2020001940. PMID 32634238
- See also: Reduced-intensity single-unit unrelated cord blood transplant with optional immune boost for nonmalignant disorders — https://pubmed.ncbi.nlm.nih.gov/32634238/